CLINICAL TRIAL: NCT01573585
Title: Effectiveness of Fast Muscle Activation and Stepping Training (FAST) on Balance and Mobility Post-stroke
Brief Title: Fast Muscle Activation and Stepping Training (FAST) Post-stroke
Acronym: FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H12-00837
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Stroke; Hemiparesis
Keywords: Physical Therapy; Exercise therapy
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): The usual care will consist of strength training, endurance, range of motion, patient education, weight shifting in standing and gait re-training.
  Interventions: Behavioral: Usual Care
- FAST protocol (Experimental): The Fast muscle activation and stepping training will be the Experimental arm of this trial. This program will be exercises emphasizing speed of movement.
  Interventions: Behavioral: FAST protocol

INTERVENTIONS:
Behavioral: Usual Care — The Usual Care program will consist of 2 sessions a week for 45 minutes for a 6 week duration.
  Arms: Usual care
Behavioral: FAST protocol — The Fast muscle activation and Stepping Training (FAST protocol) will be exercises emphasizing speed, small squats and protective steps, that will be progressed. This program will be 2 sessions a week for 45 minutes for 6 weeks in duration.
  Arms: FAST protocol

SUMMARY:
The purpose of this study is to determine whether FAST (Fast muscle Activation and Stepping Training) exercises will improve walking balance in individuals after stroke to a greater extent than usual care.

Hypothesis: The primary hypothesis is that improvements in walking balance will be larger following 12 sessions of FAST exercise retraining compared to usual care in persons in the sub-acute phase after stroke.

DETAILED DESCRIPTION:
It is estimated that 75-80% of individuals who have had a stroke will survive the acute event and be left with residual disability. Regaining independence in standing and walking is of utmost importance for patients recovering from stroke. Walking balance requires muscles in the legs and trunk to contract quickly if people lose their balance. Physical therapy plays a key role in the rehabilitation of walking balance in individuals after stroke. Given that maintaining one's balance requires fast muscle activity, rehabilitation post-stroke should focus on speed of movement. Thus we are proposing to compare a program that emphasizes speed of movement, Fast muscle Activation and Stepping Training versus an active control (usual care).

ELIGIBILITY:
Study population: Subjects with a diagnosis of stroke

Inclusion Criteria:

* first stroke (<6 months ago)
* presence of hemiparesis in the lower extremity
* minimum Berg Balance Score (BBS) of 30/56
* cognitive ability to give informed consent

Exclusion Criteria:

* bilateral stroke, or a previous stroke in the other hemisphere
* severe co-morbidity that is likely to dominate the pattern of care
* co-existing peripheral neuropathies or disorders of the vestibular apparatus
* musculoskeletal problems
* global aphasia or receptive aphasia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Community Balance and Mobility Scale | Pre treatment and Post treatment (6 weeks)

SECONDARY OUTCOMES:
Gait assessment | Pre treatment, Post treatment (6 weeks) and Retention (+1 month after treatment)
  Self selected speed and changes in electromyography
Physiological balance assessment by internal and external perturbations | Pre treatment, Post treatment (6 weeks) and Retention (+1 month after treatment)
  Electromyography and Center of pressure changes
Activities-specific Balance Confidence Scale | Pre treatment, Post treatment (6 weeks) and Retention (+1 month after treatment)
Community Balance and Mobility Scale | Post treatment and Retention (+1 month after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: S. Jayne Garland, PT, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Holy Family Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KJ, Hunt MA, Pollock CL, Bryant D, Garland SJ. Protocol for a randomized controlled clinical trial investigating the effectiveness of Fast muscle Activation and Stepping Training (FAST) for improving balance and mobility in sub-acute stroke. BMC Neurol. 2014 Oct 10;14:187. doi: 10.1186/s12883-014-0187-y. PMID 25300433
- [Derived] Peters S, Ivanova TD, Lakhani B, Boyd LA, Garland SJ. Neuroplasticity of Cortical Planning for Initiating Stepping Poststroke: A Case Series. J Neurol Phys Ther. 2020 Apr;44(2):164-172. doi: 10.1097/NPT.0000000000000311. PMID 32168159